CLINICAL TRIAL: NCT01997294
Title: Sequential Therapy of Atorvastatin Improving Tissue Reperfusion and Clinical Outcomes of ST-elevated Acute Myocardial Infarction Study（The STRAIT Study）
Brief Title: Sequential Therapy of Atorvastatin Improve Outcomes of ST-elevated Acute Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhang Qi, MD (Other)
Responsible Party: Sponsor-Investigator, Zhang Qi, MD, Visa Chief of Department of Cardiology, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RJH20130115; 2011BAI11B05 (Other Grant/Funding Number: Ministry of Science and Techology of the Pelple's Republic of China)
Record Dates: First submitted 2013-11-22; First posted 2013-11-28 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Acute Myocardial Infarction
Keywords: sequential therapy; atorvastatin; acute myocardial infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sequential therapy group (Active Comparator): 80mg atorvastatin before primary PCI (PPCI) followed by 40mg/d for 7 days after PPCI followed by 20mg/d for 1 year
  Interventions: Drug: Sequential therapy of atorvastatin
- Usual Therapy of atorvastatin (Placebo Comparator): 20mg/d before and after PPCI for 1 year
  Interventions: Drug: Sequential therapy of atorvastatin

INTERVENTIONS:
Drug: Sequential therapy of atorvastatin — 80mg atorvastatin before PPCI and 40mg/d for 7 days after PPCI

SUMMARY:
Statins have been approved to benefit patients underwent percutaneous coronary intervention (PCI). The current study is designed to evaluate the effectiveness and safety of Sequential Therapy of Atorvastatin in patients with ST-elevated myocardial infarction and receive PCI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Sighed informed consent
* Diagnosised as acute myocardial infarction
* Time frame less than 12 hours since the occurance of chest pain
* Aggred to receive sirolimus-eluted coronary stents
* Patients willing to accepte follow-up

Exclusion Criteria:

* Allegy to statins or with a history against statin therapy
* Allegy to any products that will be used during PPCI
* Disagreed to receive PPCI and other related therapy
* Existing sever liver dysfuntion that statins can not be used according to the guildlines
* Sever kidney dysfunction (creatinine >3mg/dl or eGFR<30ml/min)
* Sever left ventricular dysfunction (Killip grade 3)
* Patients are currently taking medicine that may influence the use of statin
* Patients with a history of alcohol abuse or durg abuse
* Woman during pregnancy or lactation
* Patients who has attended other clinical trials
* Patients who has received PCI or CABG previously
* Patients who can not agree to accept study protocol
* Other conditions that may not sutible for the current study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2013-01; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Events (MACE) Occourance Rate | 30 days
  1. Cardiac Death (CD)
  2. Non-fatal re-inarction (CK-MB, cTNI or cTNT elevation again and over 3 times higher than up normal limit accompanied with syptoms or EKG indication)
  3. revascularization driven by syptoms (CABG or re-PCI)

SECONDARY OUTCOMES:
Secondary Endpoints | 12 months
  1. TMP and TIMI grade chage after stents implantation; EKG ST reduction
  2. MACE ( same definition as primary endpoints)

OTHER OUTCOMES:
Safty Endpoints | 12 months
  1. Impairment of liver and kidney function
  2. Other adverse events related to statin use

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Shen, MD. PhD., Study Director — Institute of Cardiovascular Diseases, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Ruijin Hospital, Dept. of Cardiology, Shanghai, Shanghai Municipality, China